CLINICAL TRIAL: NCT02936505
Title: A Scandinavian Controlled, Randomized, Open-label, and Multi-centre Study Evaluating if Once-daily Tacrolimus or Twice-daily Cyclosporin, Reduces the 3-year Incidence of Chronic Lung Allograft Dysfunction After Lung Transplantation
Brief Title: Clinical Study Evaluating Two Treatment Protocols for Immunosuppressive Drugs. Looking at 3-year Incidence of CLAD.
Acronym: ScanCLAD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Oslo University Hospital (Other); Helsinki University Central Hospital (Other); Skane University Hospital (Other); Copenhagen University Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Göran Dellgren, MD, PhD, Vastra Gotaland Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 8.0; 154-16 (Other: EC, Gothenburg, Sweden); 2015-004137-27 (EudraCT Number); T-798-16 (amendement) (Other: EC, Gothenburg, Sweden); T002-17 (amendement) (Other: EC, Gothenburg, Sweden); T 055-18 (amendement) (Other: EC, Gothenburg, Sweden); T568-18 (amendement) (Other: EC, Gothenburg, Sweden); 2019-06057 (amendement) (Other: EC (EPM), Gothenburg, Sweden); 2021-05380-02 (amendement) (Other: EC (EPM), Gothenburg, Sweden)
Record Dates: First submitted 2016-10-15; First posted 2016-10-18 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Lung Transplantation; Allografts
Keywords: chronic lung allograft dysfunction; cyclosporin; tacrolimus; Bronchiolitis Obliterans Syndrome; Restrictive Allograft Syndrome; CLAD; immunization; renal function; survival
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Cyclosporine; Mycophenolic Acid; Antilymphocyte Serum; thymoglobulin; Adrenal Cortex Hormones; Methylprednisolone; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A:Cyclosporine (Active Comparator): Group A: Cyclosporine A, Mycophenolate mofetil (MMF) and corticosteroids according to local practice and approved label.
  Interventions: Drug: Cyclosporine; Drug: Mycophenolate mofetil (MMF); Drug: Rabbit Anti thymocyte globulin; Drug: Corticosteroids
- Arm B:Tacrolimus (Experimental): Group B: Tacrolimus (Advagraf), Mycophenolate mofetil (MMF) and corticosteroids.
  Interventions: Drug: Mycophenolate mofetil (MMF); Drug: Rabbit Anti thymocyte globulin; Drug: Corticosteroids; Drug: Tacrolimus

INTERVENTIONS:
Drug: Cyclosporine — Cyclosporin A (Sandimmun Neoral® or similar):
  * Cyclosporin A given orally pretransplant in the dose of 2-3 mg/kg.
  * Continued postop day 1 in the dose of 3mg/kgx2, according to local practice and blood concentration: 0-3 months 250-300; 3-6 months 200-250; 6-12 months 150-200; >12 months 100-150 ng/ml. Cyclosporine A will be administered twice daily.
  Other Names: Sandimmun Neural
  Arms: Arm A:Cyclosporine
Drug: Mycophenolate mofetil (MMF) — MMF target dose: 2000 mg/day (1gx2):
  o Controlled by a single Area Under the Curve (AUC) measurement day 90 with a target AUC between 40 and 60 mg.h/L and corrected accordingly.
  Other Names: Cellcept
Drug: Rabbit Anti thymocyte globulin — Induction therapy: Thymoglobulin® (Rabbit Anti thymocyte globulin)(1.5 mg/kg given immediately postoperatively).
  Other Names: Thymoglobulin®
Drug: Corticosteroids — Corticosteroids:
  * Day 0 (day of lung transplantation); 500+500mg methylprednisolone iv. before reperfusion, i.e. restoration of blood flow into the transplanted allograft.
  * From day 1: Initiated at 0.2 mg/kg/day; tapered to 0.1 mg/kg 3-6 months; less than 0,1 mg/kg > 6 months.
  Other Names: Methylprednisolon
Drug: Tacrolimus — * Tacrolimus should be given orally pretransplant in the dose of 0.1 mg/kg.
  * Continued postop day 1 according to local practice and blood concentration: 0-3 months 10-14, 3-6 months 8-12, 6-12 months 8-10, >12 months 6-8 ng/ml. Tacrolimus will be administered once daily.
  Other Names: Advagraf®
  Arms: Arm B:Tacrolimus

SUMMARY:
A controlled randomized, open-label, multi-centre study evaluating if an immunosuppressive protocol, based on ATG-induction, once daily tacrolimus-dose (Advagraf®), mycophenolate mofetil and corticosteroid reduces the incidence of chronic lung allograft dysfunction (CLAD) after lung transplantation, in comparison with a standard cyclosporin-based protocol.

DETAILED DESCRIPTION:
Study purpose:

To evaluate whether the use of a once-daily tacrolimus-dose regimen (Advagraf®), based on anti-thymocyte globulin (Thymoglobulin®) induction, mycophenolate mofetil (MMF) and corticosteroids, reduces the cumulative incidence of CLAD after de novo lung transplantation at 36 months, in comparison with a twice-daily cyclosporin-based protocol, otherwise identical between groups.

ELIGIBILITY:
Inclusion Criteria

1. Male or female lung recipients 18-70 years of age undergoing primary double (including size reduction) lung transplantation.
2. Patient willing and capable of giving written informed consent for study participation and anticipated to be able to participate in the study for 36 months.

Exclusion Criteria

1. Recipients of multiorgan transplant, and or previously transplanted with any organ, including previous lung transplantation.
2. Patients with hypersensitivity to, or other reasons to not be able to take the immunosuppressive drugs used in the study.
3. Donor lung cold ischemic time > 12 hours.
4. Patients who previously have been treated with anti-thymocyte globulin preparations (e.g. ATG-Fresenius®, Thymoglobulin®).
5. Patients who are recipients of ABO-incompatible transplants.
6. Patients with platelet count < 50,000/mm3 at the evaluation before transplantation.
7. Patients who are unlikely to comply with the study requirements.
8. Patients, and/or those receiving organs from donors, who are positive for HIV, Hepatitis B surface antigen or Hepatitis C virus.
9. Patients with donor greater than 75 years.
10. Patient who have received an unlicensed drug or therapy within one month prior to study entry or if such therapy is to be instituted post-transplantation.
11. Patient unable to participate in the study for the full 36-month period
12. Patients with any past (within the past 3-5 years) or present malignancy (other than excised basal cell carcinoma).
13. Females capable of becoming pregnant must have a negative pregnancy test prior to randomization.

Females are recommended to practice a medically approved method of birth control for the duration of the study and a period of 8 weeks following discontinuation of study medication, even where there has been a history of infertility

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with incidence of CLAD | 36 months is primary outcome
  The cumulative incidence of CLAD (including both BOS and RAS, as defined in the Appendix II) after lung transplantation.
Number of patients with incidence of CLAD | 48 months is outcome for the continuation study
  The cumulative incidence of CLAD (including both BOS and RAS, as defined by the Appendix II) at 48 months after lung transplantation.
Number of patients with incidence of CLAD | 60 months is outcome for continuation study
  The cumulative incidence of CLAD (including both BOS and RAS, as defined by the Appendix II) at 60 months after lung transplantation.
Number of patients with incidence of CLAD | 72 months is outcome for continuation study
  The cumulative incidence of CLAD (including both BOS and RAS, as defined by the Appendix II) at 72 months after lung transplantation.

SECONDARY OUTCOMES:
Glomerular Filtration Rate | 3 months
  Renal function evaluated by measured glomerular filtration rate
Primary graft dysfunction | 72 hours
  Cumulative incidence of primary graft dysfunction
Composite measure of freedom from AR, CLAD, graft and patient survival | 12 months
  Composite measure of freedom from first event of AR, CLAD, graft survival, and patient survival
Composite measure of freedom from AR, CLAD, graft and patient survival | 24 months
  Composite measure of freedom from first event of AR, CLAD, graft survival, and patient
Composite measure of freedom from AR, CLAD, graft and patient survival | 36 months
  Composite measure of freedom from first event of AR, CLAD, graft survival, and patient
Incidence of primary graft dysfunction | 72 hours
  cumulative incidence of primary graft dysfunction
Patient survival | 1 year
  Patient survival
Patient survival | 3 year
  Patient survival
Cumulative incidence of acute allograft rejection and CLAD | 6 months
  The cumulative incidence of acute allograft rejection (AR) and CLAD. - Determined by clinical criteria, computed tomography (CT) and trans bronchial lung biopsy with broncho-alveolar lavage (BAL). - Number of rejections (cellular and antibody mediated), stratified by biopsy and non-biopsy verified rejections.
Cumulative incidence of acute allograft rejection and CLAD | 1 year
  The cumulative incidence of acute allograft rejection (AR) and CLAD. - Determined by clinical criteria, computed tomography (CT) and trans bronchial lung biopsy with broncho-alveolar lavage (BAL). - Number of rejections (cellular and antibody mediated), stratified by biopsy and non-biopsy verified rejections.
Cumulative incidence of acute allograft rejection and CLAD | 3 year
  The cumulative incidence of acute allograft rejection (AR) and CLAD. - Determined by clinical criteria, computed tomography (CT) and trans bronchial lung biopsy with broncho-alveolar lavage (BAL). - Number of rejections (cellular and antibody mediated), stratified by biopsy and non-biopsy verified rejections.
Cumulative incidence of BOS and RAS | 6 months
  The cumulative incidence of BOS and RAS
Cumulative incidence of BOS and RAS | 1 year
  The cumulative incidence of BOS and RAS
Cumulative incidence of BOS and RAS | 3 year
  The cumulative incidence of BOS and RAS
Development of donor specific antibodies | 12 months
  Development of donor specific antibodies (DSA) according to specific protocol.
Development of donor specific antibodies | 24 months
  Development of donor specific antibodies (DSA) according to specific protocol.
Development of donor specific antibodies | 36 months
  Development of donor specific antibodies (DSA) according to specific protocol.
Renal function mGFR | 12 months
  Renal function evaluated by measured glomerular filtration rate (mGFR), by Iohexol or Cr-EDTA clearance.
Renal function mGFR | 24 months
  Renal function evaluated by measured glomerular filtration rate (mGFR), by Iohexol or Cr-EDTA clearance.
Renal function mGFR | 36 months
  Renal function evaluated by measured glomerular filtration rate (mGFR), by Iohexol or Cr-EDTA clearance.
Renal function cGFR | 3 months
  Renal function evaluated by calculated glomerular filtration rate (cGFR), by three different Formulas.
Renal function cGFR | 12 months
  Renal function evaluated by calculated glomerular filtration rate (cGFR), by three different Formulas.
Renal function cGFR | 24 months
  Renal function evaluated by calculated glomerular filtration rate (cGFR), by three different Formulas.
Renal function cGFR | 36 months
  Renal function evaluated by calculated glomerular filtration rate (cGFR), by three different Formulas.
Post Transplantation Diabetes Mellitus | 6 months
  The cumulative incidence of Post Transplantation Diabetes Mellitus (PTDM) after transplantation as defined below. Cumulative incidence of
  ≥2 Fasting Plasma Glucose (FPG) ≥7,0 mmol/L ≥ 30 consecutive days apart. Oral hypoglycaemic treatment ≥30 consecutive days. Insulin ≥30 consecutive days. HgbA1c ≥6.5% (according to American Diabetes Association - ADA)Symptoms of Diabetes and Random Plasma Glucose (RPG) ≥ 11.1 mmol/L.
  2-hour Plasma Glucose (2-hPG) ≥ 11.1 mmol/L during an oral glucose tolerance test (OGTT). Baseline OGTT will be performed pre-transplant.
Post Transplantation Diabetes Mellitus | 12 months
  The cumulative incidence of Post Transplantation Diabetes Mellitus (PTDM) after transplantation as defined below. Cumulative incidence of
  ≥2 Fasting Plasma Glucose (FPG) ≥7,0 mmol/L ≥ 30 consecutive days apart. Oral hypoglycaemic treatment ≥30 consecutive days. Insulin ≥30 consecutive days. HgbA1c ≥6.5% (according to American Diabetes Association - ADA) Symptoms of Diabetes and Random Plasma Glucose (RPG) ≥ 11.1 mmol/L. 2-hour Plasma Glucose (2-hPG) ≥ 11.1 mmol/L during an oral glucose tolerance test (OGTT). Baseline OGTT will be performed pre-transplant.
Post Transplantation Diabetes Mellitus | 24 months
  The cumulative incidence of Post Transplantation Diabetes Mellitus (PTDM) after transplantation as defined below. Cumulative incidence of
  ≥2 Fasting Plasma Glucose (FPG) ≥7,0 mmol/L ≥ 30 consecutive days apart. Oral hypoglycaemic treatment ≥30 consecutive days. Insulin ≥30 consecutive days. HgbA1c ≥6.5% (according to American Diabetes Association - ADA) Symptoms of Diabetes and Random Plasma Glucose (RPG) ≥ 11.1 mmol/L. 2-hour Plasma Glucose (2-hPG) ≥ 11.1 mmol/L during an oral glucose tolerance test (OGTT). Baseline OGTT will be performed pre-transplant.
Post Transplantation Diabetes Mellitus | 36 months
  The cumulative incidence of Post Transplantation Diabetes Mellitus (PTDM) after transplantation as defined below -Cumulative incidence of:
  ≥2 Fasting Plasma Glucose (FPG) ≥7,0 mmol/L ≥ 30 consecutive days apart. Oral hypoglycaemic treatment ≥30 consecutive days. Insulin ≥30 consecutive days. HgbA1c ≥6.5% (according to American Diabetes Association - ADA)Symptoms of Diabetes and Random Plasma Glucose (RPG) ≥ 11.1 mmol/L.
  2-hour Plasma Glucose (2-hPG) ≥ 11.1 mmol/L during an oral glucose tolerance test (OGTT). Baseline OGTT will be performed pre-transplant.
Antidiabetic medication | 6 months
  Use of antidiabetic medication
Antidiabetic medication | 12 months
  Use of antidiabetic medication
Antidiabetic medication | 24 months
  Use of antidiabetic medication
Antidiabetic medication | 36 months
  Use of antidiabetic medication
Antihypertensive and lipid lowering drugs | 12 months
  Incidence and number of antihypertensive and lipid lowering drug
Antihypertensive and lipid lowering drugs | 24 months
  Incidence and number of antihypertensive and lipid lowering drug
Antihypertensive and lipid lowering drugs | 36 months
  Incidence and number of antihypertensive and lipid lowering drug
Proteinuria | 12 months
  Development and magnitude of proteinuria
Proteinuria | 24 months
  Development and magnitude of proteinuria
Proteinuria | 36 months
  Development and magnitude of proteinuria
Lipid profile | 12 months
  Lipid profile (Total cholesterol, LDL-cholesterol, HDL-cholesterol, Triglycerides, TSH, T4, HbA1c)
Lipid profile | 24 months
  Lipid profile (Total cholesterol, LDL-cholesterol, HDL-cholesterol, Triglycerides, TSH, T4, HbA1c)
Lipid profile | 36 months
  Lipid profile (Total cholesterol, LDL-cholesterol, HDL-cholesterol, Triglycerides, TSH, T4, HbA1c)
Cytomegalovirus | 0-36 months
  Incidence of Cytomegalovirus (CMV) that required treatment (CMV-infection and CMV syndrome).
Malignancy stratified by post-transplant lymphoproliferative disorder (PTLD) and all other cancers. | 36 months
  Cumulative incidence of malignancy stratified by post-transplant lymphoproliferative disorder (PTLD) and all other cancers.
Safety and tolerability | 0-36 months
  Safety and tolerability
Quality of life assessed by EQ5D Questionnaire | 12 months
  Quality of life, the relative difference over time will be investigated after LTx, where 5 questions are raised and answer is between 11111 (no problems) and 33333 (extreme problems in all dimensions)
Quality of life assessed by St Georges Respiratory Questionnaire (SGRQ) | 12 months
  Quality of life, the relative difference over time will be investigated after LTx. The SGRQ total score ranges from 0 to 100 where 100 indicates the worst quality of life.
Quality of life, assessed by EQ5D Questionnaire | 24 months
  Quality of life, the relative difference over time will be investigated after LTx, where 5 questions are raised and answer is between 11111 (no problems) and 33333 (extreme problems in all dimensions).
Quality of life, assessed by St Georges Respiratory Questionnaire (SGRQ) | 24 months
  Quality of life, the relative difference over time will be investigated after LTx. The SGRQ total score ranges from 0 to 100 where 100 indicates the worst quality of life.
Quality of life, assessed by EQ5D Questionnaire (SGRQ) | 36 months
  Quality of life, the relative difference over time will be investigated after LTx, where 5 questions are raised and answer is between 11111 (no problems) and 33333 (extreme problems in all dimensions).
Quality of life, assessed by St Georges Respiratory Questionnaire (SGRQ) | 36 months
  Quality of life, the relative difference over time will be investigated after LTx. The SGRQ total score ranges from 0 to 100 where 100 indicates the worst quality of life.
Pharmacokinetics, of the Tacrolimus drug in patients in the CF sub group population | week 4
  Define the pharmacokinetics from whole blood concentrations at 0h after administration, of Tacrolimus in non-CF patients (n=12) and all included CF patients (n=15-20) undergoing primary lung transplantation (LTx) treated with an Advagraf® based-immunosuppression.
Pharmacokinetics, of the Tacrolimus drug in patients in the CF sub group population | week 4
  Define the pharmacokinetics from whole blood concentrations at 1h after administration of Tacrolimus in non-CF patients (n=12) and all included CF patients (n=15-20) undergoing primary lung transplantation (LTx) treated with an Advagraf® based-immunosuppression.
Pharmacokinetics, of the Tacrolimus drug in patients in the CF sub group population | week 4
  Define the pharmacokinetics from whole blood concentrations at 2h after administration of Tacrolimus in non-CF patients (n=12) and all included CF patients (n=15-20) undergoing primary lung transplantation (LTx) treated with an Advagraf® based-immunosuppression.
Pharmacokinetics, of the Tacrolimus drug in patients in the CF sub group population | week 4
  Define the pharmacokinetics from whole blood concentrations at 3h after administration of Tacrolimus in non-CF patients (n=12) and all included CF patients (n=15-20) undergoing primary lung transplantation (LTx) treated with an Advagraf® based-immunosuppression.
Pharmacokinetics, of the Tacrolimus drug in patients in the CF sub group population | week 4
  Define the pharmacokinetics from whole blood concentrations at 4h after administration of Tacrolimus in non-CF patients (n=12) and all included CF patients (n=15-20) undergoing primary lung transplantation (LTx) treated with an Advagraf® based-immunosuppression.
Pharmacokinetics, of the Tacrolimus drug in patients in the CF sub group population | week 4
  Define the pharmacokinetics from whole blood concentrations at 6h after administration of Tacrolimus in non-CF patients (n=12) and all included CF patients (n=15-20) undergoing primary lung transplantation (LTx) treated with an Advagraf® based-immunosuppression.
Pharmacokinetics, of the Tacrolimus drug in patients in the CF sub group population | week 4
  Define the pharmacokinetics (from whole blood concentrations from at 8h after administration and of Tacrolimus in non-CF patients (n=12) and all included CF patients (n=15-20) undergoing primary lung transplantation (LTx) treated with an Advagraf® based-immunosuppression.
Pharmacokinetics, of the Tacrolimus drug in patients in the CF sub group population | week 4
  Define the pharmacokinetics (from whole blood concentrations from at 10h after administration and of Tacrolimus in non-CF patients (n=12) and all included CF patients (n=15-20) undergoing primary lung transplantation (LTx) treated with an Advagraf® based-immunosuppression.
Pharmacokinetics, of the Tacrolimus drug in patients in the CF sub group population | week 4
  Define the pharmacokinetics (from whole blood concentrations at 12h after administration and of Tacrolimus in non-CF patients (n=12) and all included CF patients (n=15-20) undergoing primary lung transplantation (LTx) treated with an Advagraf® based-immunosuppression.
Pharmacokinetics, of the Tacrolimus drug in patients in the CF sub group population | week 4
  Define the pharmacokinetics from whole blood concentrations at 23h after administration and of Tacrolimus in non-CF patients (n=12) and all included CF patients (n=15-20) undergoing primary lung transplantation (LTx) treated with an Advagraf® based-immunosuppression.
Pharmacokinetics, of the Tacrolimus drug in patients in the CF sub group population | week 4
  Define the pharmacokinetics from whole blood concentrations at 24h after administration and of Tacrolimus in non-CF patients (n=12) and all included CF patients (n=15-20) undergoing primary lung transplantation (LTx) treated with an Advagraf® based-immunosuppression.
Pharmacokinetics, of the Tacrolimus drug in patients in the CF sub group population | week 4
  Define the pharmacokinetics as an AUC construction, of Tacrolimus in non-CF patients (n=12) and all included CF patients (n=15-20) undergoing primary lung transplantation (LTx) treated with an Advagraf® based-immunosuppression.
Pharmacokinetics of the Tacrolimus drug in patients in the CF sub group | 6 months
  Define the pharmacokinetics as an AUC construction, of Tacrolimus in non-CF patients (n=12) and all included CF patients (n=15-20) undergoing primary lung transplantation (LTx) treated with an Advagraf® based-immunosuppression.
Immunological equipotency of tacrolimus and cyclosporine A | 0-36 months
  Immunological equipotency of tacrolimus once daily (OD) and cyclosporine A twice daily (BiD) in vivo and in vitro, according to separate protocol.
Occurrence of treatment failures | 0-36 months
  Occurrence of treatment failures up to or at 36 months; defined as a composite endpoint of graft loss, death, loss to follow up or discontinuation due to lack of efficacy or toxicity (at least one condition must be present).
Recovery of right heart function | 0-36 months
  Recovery of right heart function irrespective of diagnosis in patients with pulmonary arterial hypertension (PAH, categories 1-5 according to WHO 1-5).

CONTACTS AND LOCATIONS:
Overall Officials: Göran Dellgren, MD, PhD, Study Chair — Sahlgrenska Univ Hospital
Locations (5):
- Rigshospitalet, Copenhagen, Denmark
- Helsinki University Hospital, Helsinki, Finland
- Oslo University Hospital, Oslo, Norway
- Sweden (2):
  - Sahlgrenska Univ Hospital, Gothenburg
  - Skåne University Hospital, Lund

IPD SHARING:
Plan to Share IPD: No
Potentially this can be done, but needs to be according to GDPR. Figures with pulmonary function tests over time and related to CLAD are constructed in the study.

REFERENCES:
- [Background] Dellgren G, Lund TK, Raivio P, Leuckfeld I, Svahn J, Magnusson J, Riise GC. Design and Rationale of a Scandinavian Multicenter Randomized Study Evaluating if Once-Daily Tacrolimus Versus Twice-Daily Cyclosporine Reduces the 3-year Incidence of Chronic Lung Allograft Dysfunction After Lung Transplantation (ScanCLAD Study). Adv Ther. 2020 Mar;37(3):1260-1275. doi: 10.1007/s12325-020-01224-1. Epub 2020 Jan 28. PMID 31993943
- [Derived] Dellgren G, Lund TK, Raivio P, Leuckfeld I, Svahn J, Holmberg EC, Olsen PS, Halme M, Fiane A, Lindstedt S, Riise GC, Magnusson J. Effect of once-per-day tacrolimus versus twice-per-day ciclosporin on 3-year incidence of chronic lung allograft dysfunction after lung transplantation in Scandinavia (ScanCLAD): a multicentre randomised controlled trial. Lancet Respir Med. 2024 Jan;12(1):34-44. doi: 10.1016/S2213-2600(23)00293-X. Epub 2023 Sep 10. PMID 37703908
- See also: Design manuscript — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7089723/